CLINICAL TRIAL: NCT06734910
Title: Effectiveness of a Digital Support Intervention (HealthyPregnancy) for Pregnant Women with a BMI At 25 or Above (BMI≥25) in Addition to Standard Care: a Stepped-wedge Cluster Randomized Controlled Trial
Brief Title: HealthyPregnancy - Digital Support for Pregnant Women with a BMI At 25 or Above (BMI≥25)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Clinical Research and Prevention (Network)
Collaborators: Nordsjaellands Hospital (Other); Slagelse Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: R232-A5142
Record Dates: First submitted 2024-11-25; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy Related; Weight Gain
Keywords: Pregnancy; Gestational weight gain; Mental well-being; Digital interventions; Physical activity; Diet
MeSH Terms: conditions — Weight Gain; Gestational Weight Gain; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomization of two study sites in three steps:
  Step 1: Both study sites acting as control. Step 2: One study site acting as control, 1 study site acting as intervention. Step 3: Both study sites acting as intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Standard antenatal care.
- HealthyPregnancy group (Active Comparator): Digital care guide as supplement to standard antenatal care.
  Interventions: Behavioral: HealthyPregnancy

INTERVENTIONS:
Behavioral: HealthyPregnancy — A digital care guide comprising of:
  1. Information about diet, exercise and mental wellbeing in pregnancy. Presented in text, video and audio material featuring various healthcare professionals.
  2. Online exercise. Access to live online structured physical exercise twice a week and to an off line library of exercise videos.
  3. Chat function with possibility to chat safely with healthcare professionals.
  4. Push-notifications reminding the participants of upcoming antenatal appointments.
  In addition an invitation to monthly café sessions focusing on e.g., mental health, parenting skills, breastfeeding and healthy lifestyle.
  Arms: HealthyPregnancy group

SUMMARY:
The study aims to examine the effectiveness of a digital care guide offering support and information on diet, physical exercise and mental well-being on pregnancy weight gain among pregnant women with a BMI at 25 or above in a stepped-wedge cluster randomised study.

The investigators hypothesise that access to a digital care guide focusing on diet, exercise and mental support, will support a reduced weight gain in pregnancy and improve the mental wellbeing of the participants.

DETAILED DESCRIPTION:
Being overweight is the most prevailing health issue among women of reproductive age, and in Denmark, the proportion of pregnant women with a body mass index at or above 25 (BMI≥25) is nearing 40%.

Women with overweight are at increased risk of complications in pregnancy and labor such as hypertensive disorders, gestational diabetes (GDM), and Cesarean section. Children of women with overweight more often have a high birthweight and are less likely to be breastfed, than children of women with a normal BMI. Both women and offspring, face an increased risk of overweight or obesity later in life. The risk of complications can increase if the pregnant woman gains excessive weight during pregnancy and conversely, reducing pregnancy weight gain can lower the risk of complications. However, more than half (60%) of pregnant women with overweight do not adhere to the pregnancy weight gain recommendations. In addition, only around one third of pregnant women with overweight meet the recommended daily levels of physical activity. This emphasizes a significant potential for prevention strategies focused on promoting healthy weight gain and physical activity during pregnancy.

It has previously been established, that interventions focusing on physical activity and nutritional counselling can help women with overweight reduce excessive pregnancy weight gain. However, traditional lifestyle interventions can be both cost-intensive and resource-demanding to implement. With digital technologies, lifestyle interventions have potential to less resource-intensive testing and implementation. New research indicates that a digital application with information on a healthy diet and physical activity may have potential to help women with overweight reduce pregnancy weight gain.

At Nordsjaellands Hospital and Slagelse Hospital respectively 37% and 49% of pregnant women are overweight with a BMI≥25. Pregnant women with overweight are offered standard care at Slagelse Hospital and at Nordsjaellands Hospital women with a BMI above 35 receive a minor supplement to standard care. However, both pregnant women and healthcare professionals request tailored and evidence-based care.

The aim of the HealthyPregnancy study is to evaluate the effect of a digital care guide offering support and information on diet, physical exercise, and mental well-being on gestational weight gain. The digital care guide will be tested in a stepped wedge cluster randomized controlled trial including 450 pregnant women with a BMI at 25 or above.

A secondary aim is to evaluate the effect of the digital care guide on pregnancy and diabetes outcomes among participating women diagnosed with gestational diabetes.

HealthyPregnancy is carried out in collaboration between Center for Clinical Research and Prevention, Nordsjaellands Hospital and Slagelse Hospital.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 or above at first prenatal visit
* Age 18 years or older
* Singleton pregnancy
* Appropriate Danish or English language skills
* Written informed consent

Exclusion Criteria:

* Age under 18 years
* Multiple pregnancy
* Gestational age above 16+0 at inclusion
* Alcohol or drug abuse
* Being diagnosed with eating disorder, schizophrenia, psychosis, or similar
* Diagnosis of malformations or chromosomal disorder in the fetus
* Conditions that lead to recommendations against physical activity during pregnancy e.g., cerclage.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Gestational weight gain | At inclusion and delivery
  Weight gain during pregnancy in kilograms

SECONDARY OUTCOMES:
Postpartum weight retention | Eight weeks after delivery and one year after delivery.
  Self-reported weight in kilograms
Mental well-being | At inclusion, gestational week 35-37, eight weeks after delivery and one year after delivery.
  Mental well-being is measured with the "World Health Organisation Five Well-being Index" (WHO-5). The lowest score of the scale is 0 and the highest total score is 100. Higher scores indicating better mental well-being.
Symptoms of depression | At inclusion, gestational week 35-37, eight weeks after delivery and one year after delivery.
  Symptoms of depression are measured with the "Edinburgh Postnatal Depression Scale" (EPDS) will be defined as cutoff score ≥ 13 and a cutoff score ≥ 10. The scale measures the intensity of common depressive symptoms on a 4-point Likert scale (0-3), where 0 indicates absence of depressive symptoms and 3 indicates the highest amount of depressive symptoms. The lowest score of the scale is 0 and the highest total score is 30.
Functional ability | At inclusion, gestational week 35-37, eight weeks after delivery and one year after delivery.
  Functional ability is measured with the "12-item General Health Questionnaire" (GHQ-12). The GHQ-12 consists of 12 items, with total scores ranging from 0 to 36, with higher scores indicating higher levels of psychological distress.
Digital health competence | At inclusion, gestational week 35-37
  Digital health competence is measured with the "eHealth Literacy Questionnaire" (eHLQ), using subscales 1. Using technology to process health information, 3. Ability to actively engage with digital services and 5. Motivated to engage in digital services.
  Each subscale is scored individually and no overall eHLQ score is calculated. Subscales consists of 4 to 6 items on a 4-point Likert scale ranging from "strongly disagree" to "strongly agree", and higher scores indicate higher abilities
Maternal sleep | At inclusion, gestational week 35-37 and one year after delivery.
  Maternal sleep quality is measured with the "Pittsburgh Sleep Quality Index" (PSQI). The global score range from 0-21 with higher scores indicating worse sleep quality.
Exercise self-efficacy | At inclusion, gestational week 35-37, eight weeks after delivery and one year after delivery.
  Exercise self-efficacy is measured with the Danish version of the "Pregnancy Exercise Self-Efficacy Scale" (P-ESES-DK). The total score of the scale range from 10 to 50, with higher scores indicating higher self-efficacy.
Physical activity in pregnancy | At inclusion, gestational week 35-37, eight weeks after delivery and one year after delivery.
  Physical activity in pregnancy is subjectively measured with the Danish version of the "Pregnancy Physical Activity Questionnaire" (PPAQ-DK).
Pregnancy complications | 2 weeks post partum
  Diagnosis with gestational diabetes, pregnancy induced hypertension or preeclampsia during pregnancy
Sick leave in pregnancy | At inclusion, gestational week 35-37.
  Percentage of participants with sick leave, no matter cause. Sick leave will be measured in days
Antenatal contacts | 2 weeks post partum
  Antenatal contacts measured as number of scheduled and unscheduled visits with obstetric doctors and midwifes
Pregnancy length | 2 weeks post partum
  Gestational age at delivery.
Onset of labor | 2 weeks post partum
  Onset of labor will be measured with spontaneous onset of labor or induced labor respectively (n/%).
Use of epidural analgesia | 2 weeks post partum
  Use of epidural analgesia will be measured by yes or no (n/%).
Use of oxytocin for augmentation during labor | 2 weeks post partum
  Use of oxytocin for augmentation during labor will be measured by yes or no (n/%).
Treatment with antibiotics during labor | 2 weeks post partum
  Treatment with antibiotics during labor will be measured by yes or no (n/%).
Mode of delivery | 2 weeks post partum
  Mode of delivery will be measured with spontaneous vaginal, instrumental vaginal or Caesarean section respectively (n/%).
Duration of labor | 2 weeks post partum
  Duration of labor will be measured by hours of active labor.
Shoulder dystocia | 2 weeks post partum
  Shoulder dystocia will be measured as yes or no (n/%).
Postpartum hemorrhage | 2 weeks post partum
  Postpartum hemorrhage is measured as hemorrhage at or above 1000 ml yes or no (n/%).
Birth weight | 2 weeks post partum
  Birth weight will be measured in kilograms (mean and SD).
Newborn's well-being at time of delivery (Apgar score) | Delivery
  Newborn's well-being at time of delivery will be measured by Apgar score (yes or no to an Apgar score ≤ 7 at 5 minutes postpartum) (n/%).
Newborn's well-being at time of delivery (pH-value in cord blood) | Delivery
  Newborn's well-being at time of delivery will be measured by the pH-value in the cord blood at time of delivery.
Admittance to neonatal intensive care unit in relation to delivery | 2 weeks post partum
  Admittance to neonatal intensive care unit in relation to delivery is measured as yes or no (n/%).
Neonatal re-admittance | 2 weeks post partum
  Neonatal re-admittance is measured as yes or no to hospital admittance within the first two weeks after initial discharge (mature infants only).
Hospitalization, length of stay | 2 weeks post partum
  The duration of hospitalization will be measured in days.
Breastfeeding intention | Gestational week 35-37, eight weeks after delivery and one year after delivery.
  Self-reported breastfeeding intention is measured with yes or no (n/%).
Intended duration of breastfeeding | Gestational week 35-37, eight weeks after delivery and one year after delivery.
  Self-reported intended duration of breastfeeding intention is measured in months.
Breastfeeding duration | Gestational week 35-37, eight weeks after delivery and one year after delivery.
  Self-reported duration of full and partial breastfeeding respectively is measured in months.
Postpartum oral glucose tolerance test | One year postpartum
  Postpartum oral glucose tolerance test is measured as yes or no (only women diagnosed with gestational diabetes).
Self-reported blood glucose values | 2 weeks post partum
  Self-reported blood glucose values during pregnancy are measured in mmol/l (only women diagnosed with gestational diabetes).
Treatment with insulin during pregnancy | 2 weeks post partum
  Treatment with insulin during pregnancy are measured with yes or no (only women diagnosed with gestational diabetes).

OTHER OUTCOMES:
Diet quality | Baseline, gestational week 35-37, eight weeks after delivery and one year after delivery.
  Self-rated diet quality will be measured by percentage of participants in each of five categories of diet quality (very healthy, healthy, somewhat healthy, unhealthy, very unhealthy).
Diet | Baseline, gestational week 35-37, eight weeks after delivery and one year after delivery.
  Diet will be measured by self-reported frequency of 20 selected foods and drinks (more than once daily, 5-7 times a week, 3-4 times a week, 1-2 times a week, rarely/never). Exploratory outcome.
Body composition | Gestational age 35-37
  Body composition during pregnancy, determined as the ratio of fatty mass to lean mass, are measured with BodPod using a Air Displacement Plethysmography System (only a sub-sample of women recrutied at NOH).
Use of the HealthyPregnancy digital application | 2 weeks post partum
  Use of the HealthyPregnancy digital application is measured as the percentages of women within three categories of engagement (low engagement, medium engagement, high engagement). Engagement data is available from the platform Emento in which the HealthyPregnancy digital application is embedded.
Prenatal caregiving expectations | Gestational week 35-37
  Prenatal caregiving expectations are measured with the"Prenatal Caregiving Expectations Questionnaire - Revised version" (PCEQ-R). Percentages of women with helpless-dysregulated, anxious-hyperactivated, and avoidant-deactivated caregiving representations respectively.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Nordsjaellands Hospital, Hillerød
  - Slagelse Hospital, Slagelse

IPD SHARING:
Plan to Share IPD: Undecided
Undecided: It is not yet known if there will be a plan to make IPD available.